CLINICAL TRIAL: NCT01696162
Title: Conventional Home Exercise Programs Versus Electronic Home Exercise Versus Artificial Intelligence "Virtual Therapy" for Anterior Knee Pain: a Prospective Randomized Comparative Trial.
Brief Title: Conventional Home Exercise Programs Versus Electronic Home Exercise Versus Artificial Intelligence "Virtual Therapy" for Anterior Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simpletherapy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 413
Record Dates: First submitted 2012-09-15; First posted 2012-09-28 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Knee pain; Anterior knee pain; Patellofemoral; Patellofemoral syndrome; Runners knee
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PDF exercise sheets (Active Comparator): Participants in this arm will receive a PDF sheet of 6 exercises that are commonly administered for the treatment of anterior knee pain. They will be asked to perform the exercises three times a week for 6 weeks. A questionnaire will be administered at the three, six and twelve week mark to evaluate efficacy, compliance and safety.
  Interventions: Other: PDF Exercise Sheets
- Limited Exercise Videos (Active Comparator): Participants in this arm will receive the same six exercises as provided in the PDF sheet in arm 1 in a video format. They will be asked to perform the exercises three times per week for 6 weeks.
  A questionnaire will be administered at the three, six and twelve week mark to evaluate efficacy, compliance and safety.
  Interventions: Other: Limited Exercise Videos
- Algorithm based Exercise Videos (Experimental): Participants in this arm will be provided a 6 week regimen of exercise videos for their anterior knee pain. Following each exercise session, the participant will be asked for their input concerning each exercise. The algorithm will adjust the exercise regimen for the next session based on the participants input. A questionnaire will be administered at the three, six and twelve week mark to evaluate efficacy, compliance and safety.
  Interventions: Other: Algorithm based Exercise Videos

INTERVENTIONS:
Other: Algorithm based Exercise Videos — The algorithm will adjust the exercises in each session based upon the participant's feedback.
  Arms: Algorithm based Exercise Videos
Other: PDF Exercise Sheets — A sheet of six exercises with descriptions on how to perform them properly
  Arms: PDF exercise sheets
Other: Limited Exercise Videos — Video of 6 exercises that provide instruction on how to perform the exercises
  Arms: Limited Exercise Videos

SUMMARY:
This is a clinical research trial to evaluate the efficacy of delivering exercise therapy for knee pain via the Internet utilizing an algorithm designed to adjust a home exercise program based on user input. The investigators hypothesize that exercise therapy can be delivered safely and effectively with increased participant satisfaction compared to the current standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 with anterior knee pain
* Have computer access
* Cleared for exercise by a medical professional, if not possible or a medical professional on the study team over the phone and the PAR-Q (Physical Activity Readiness Questionnaire)
* Have consented to participate in the trial

Exclusion Criteria:

* Age < 18 or > 64
* Screened as unsafe for exercise by a medical professional or the, study team and/ or Screened out by the PAR-Q
* Does not consent to the trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The 3 and 6 week survey data evaluating efficacy of the algorithm | 6 months
  Each participant will be asked at the 3, 6 and 12 week mark to fill out a survey questionnaire that evaluates their knee pain to determine if their knee pain has improved.

SECONDARY OUTCOMES:
Participant compliance | 6 months
  We will ask the participant at the 3, 6 and 12 week mark questions concerning whether they enjoyed the video exercises and whether they would do them again.
Safety | 6 months
  The screening questionnaires will be evaluated for their safety and efficacy. This will be evaluated by having followup at the 3, 6 and 12 week marks and asking if the participant had any adverse event either via phone calls or survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Garino, MD, Principal Investigator — Simpletherapy
Locations (1):
- Simpletherapy, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Baker KR, Nelson ME, Felson DT, Layne JE, Sarno R, Roubenoff R. The efficacy of home based progressive strength training in older adults with knee osteoarthritis: a randomized controlled trial. J Rheumatol. 2001 Jul;28(7):1655-65. PMID 11469475
- [Background] Margolis SA, Paule RC, Ziegler RG. Ascorbic and dehydroascorbic acids measured in plasma preserved with dithiothreitol or metaphosphoric acid. Clin Chem. 1990 Oct;36(10):1750-5. PMID 2208649
- [Background] Bassett SF, Prapavessis H. Home-based physical therapy intervention with adherence-enhancing strategies versus clinic-based management for patients with ankle sprains. Phys Ther. 2007 Sep;87(9):1132-43. doi: 10.2522/ptj.20060260. Epub 2007 Jul 3. PMID 17609331
- [Background] Crossley K, Bennell K, Green S, Cowan S, McConnell J. Physical therapy for patellofemoral pain: a randomized, double-blinded, placebo-controlled trial. Am J Sports Med. 2002 Nov-Dec;30(6):857-65. doi: 10.1177/03635465020300061701. PMID 12435653
- [Derived] Kim TWB, Gay N, Khemka A, Garino J. Internet-Based Exercise Therapy Using Algorithms for Conservative Treatment of Anterior Knee Pain: A Pragmatic Randomized Controlled Trial. JMIR Rehabil Assist Technol. 2016 Dec 14;3(2):e12. doi: 10.2196/rehab.5148. PMID 28582256
- See also: Trial Enrollment Webpage — http://www.simpletherapy.com/how-simpletherapy-works/